CLINICAL TRIAL: NCT01741961
Title: 4-year Follow-up After Ahmed Glaucoma Valve Implantation for Lowering Intraocular Pressure in Different Types of Glaucoma
Brief Title: Long Term Outcome After Ahmed Glaucoma Valve
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Karin Pillunat, Principal Investigator, Technische Universität Dresden
Other Study IDs: Ahmed-LTO
Record Dates: First submitted 2012-11-22; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Glaucoma
Keywords: uncontrolled glaucoma; glaucoma drainage device
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- glaucoma, surgery, Ahmed valve: Patients with uncontrolled glaucoma undergoing Ahmed glaucoma valve implantation for intraocular pressure reduction.
  Interventions: Procedure: Ahmed valve

INTERVENTIONS:
Procedure: Ahmed valve — The flexible plate 7 (FP7) model (New World Medical) was implanted in patients with uncontrolled glaucoma.

SUMMARY:
Long term results after Ahmed glaucoma valve implantation for uncontrolled glaucoma are retrospectively examined.

DETAILED DESCRIPTION:
The development of intraocular pressure, visual acuity, number of glaucoma medication, number of complications and necessity of revision operations after Ahmed glaucoma valve implantation for uncontrolled glaucoma is examined yearly for a period of 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from medically uncontrolled glaucoma
* Informed consent

Exclusion Criteria:

* healthy subjects
* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from uncontrolled glaucoma, most often after multiple ocular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2006-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
intraocular pressure reduction | 4 years
  The reduction of intraocular pressure after Ahmed glaucoma valve implantation is observed over a period of 4 years.

SECONDARY OUTCOMES:
development of visual acuity | 4 years
  The development of visual acuity after Ahmed glaucoma valve implantation is being examined over a period of 4 years.

OTHER OUTCOMES:
reduction of glaucoma medication | 4 years
  The number of glaucoma medication after Ahmed glaucoma valve implantation are being examined over a period of 4 years.
postoperative complications | 4 years
  Possible postoperative complications after Ahmed glaucoma valve implantation are being examined over a period of 4 years.
need for revision operation | 4 years
  The need for revision operations after Ahmed glaucoma valve implantation is being examined over a period of 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Karin R Pillunat, MD, Principal Investigator — University Dresden, Eye Clinic
Locations (1):
- University Eye Clinic Dresden, Dresden, Saxony, Germany